CLINICAL TRIAL: NCT03542799
Title: Phase I/II Study of EGFR-IL12-CART Cells for Patients With Metastatic Colorectal Cancer
Brief Title: EGFR-IL12-CART Cells for Patients With Metastatic Colorectal Cancer
Acronym: EGFRCART
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Collaborators: The Pregene (ShenZhen) Biotechnology Company, Ltd. (Industry)
Responsible Party: Principal Investigator, tiangeng, Chief physician, Shenzhen Second People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol. PGCAR/EGFR012
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 (Experimental): anti-tumor response of EGFR IL12 CART
  Interventions: Biological: EGFR IL12 CART

INTERVENTIONS:
Biological: EGFR IL12 CART — EGFR IL12 CART cells will be administered using a split dose on day0 (10%),1(30%), and 2(60%)

SUMMARY:
This is a clinical study to observe the maximum tolerated dose (MTD) and the safety and feasibility of chimeric antigen receptor EGFR (EGFR -IL12 -CART) cells in metastatic patients with colorectal cancer.

DETAILED DESCRIPTION:
This is a study for the patients with colorectal cancer. Maximum tolerated dose climbing test is expected into the group of 9 cases of patients. And Phase II expected into the group of 11 subjects, selected the above safe dose, carrying out a research into the clinical effectiveness. Subjects will be collected their T cells and modify them, the modification is a genetic change, that EGFR:4-1BB:CD28:CD3 modified T cells, in order to tells the T cells to recognize their target tumor cells and potentially kill them, but not other normal cells in the subject's body. The CART cells will then be expanded in vitro and then administered to subjects. Fourth generation CART, also known as TRUCKs (T cells redirected for universal cytokine before), mainly in order to improve the effect of solid tumor treatment and design, through NFAT transcription factors inducing expression of IL - 12, overcome the solid tumor within the tumor microenvironment of CART limit the function of cellsThe purpose of this study is observe the MTD and to assess the safety and feasibility of CART cells in the patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years to 70 years;
2. Clinical diagnosis of EGFR positive for patients with metastatic colorectal cancer;
3. Patients must have a KPS of >80, expected survival > 3 months;
4. Patients must have at least one measurable lesions;
5. Recently did not use glucocorticoid;
6. Patients must have evidence of adequate hepatic and renal function as evidenced by the following laboratory parameters: WBC ≥ 3.0×109/L, Hb ≥90 g/L, PLT ≥100×109/L）; AST ≤2.5ULN，ALT ≤ 2.5ULN; Cr≤ 3ULN; TBIL≤ 3ULN，
7. Patients must have a good heart function (LVEF>50%) ;
8. Patients must be willing to practice birth control during and for three months following treatment.NOTE:female participants of reproductive potential must have a negative serum pregnancy test, and willing to practice birth control during and for three months following treatment；
9. Patients must be willing to sign an informed consent.

Exclusion Criteria:

1. Patients with other cancer history;
2. Patients allergic to cetuximab;
3. Patients with severe bronchitis, bronchial asthma, or severs pneumonia;
4. Patients with uncontrolled active infections (bacteria, viruses or fungi infection) ;
5. Patients with acute and chronic GVHD (graft versus host disease)
6. Patients with severe autoimmune diseases;
7. Previously treatment with T cell inhibitors (cyclophosphamide, FK506);
8. Patients with active hepatitis B or hepatitis C infection, HIV infection, syphilis serology reaction positive;
9. Patients who are participating or participated any other clinical research in the past 1 months;
10. Pregnant and/or lactating women will be excluded; -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-22 (Estimated); Primary Completion 2020-05-23 (Estimated); Study Completion 2021-05-23 (Estimated)

PRIMARY OUTCOMES:
Safety: Occurrence of study related adverse events | 24 weeks
  Occurrence of study related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Effectiveness: Changes of tumor markers | 24 weeks
  Changes of tumor markers CA-199, AFP and CEA
Effectiveness: duration of in vivo survival of EGFR CART | 1 year
  Determine duration of in vivo survival of EGFR CART

CONTACTS AND LOCATIONS:
Locations (1):
- Geng Tian 13724395569 Tiangeng666@Aliyun.Com, Shenzhen, GuangGong, China

IPD SHARING:
Plan to Share IPD: No